CLINICAL TRIAL: NCT01485601
Title: A Randomised, Double-blind, Multi-centre, Phase II, Optimal Dose-finding Study to Determine the Safety and Efficacy of MT10109 (Clostridium Botulinum Toxin Type A) in Subjects With Moderate to Severe Glabellar Lines in Comparison to BOTOX®
Brief Title: Safety and Efficacy Study of Botulinum Toxin Type A to Treat Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-GPRT-GL01
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-07

CONDITIONS: Glabellar Frown Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MT10109 (Experimental): Clostridium botulinum toxin type A
  Interventions: Biological: MT10109
- Botox (registered trade mark) (Active Comparator): Clostridium botulinum toxin type A
  Interventions: Biological: MT10109

INTERVENTIONS:
Biological: MT10109 — Single dose intramuscular injection MT10109 vs Botox®

SUMMARY:
The purpose of this study is to find an optimal dose to determine the safety and tolerability of a single dose of MT10109(clostridium botulinum type A) administered by intramuscular injection in subjects with glabellar lines compared with the standard dose of BOTOX®

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 75 years with glabellar facial lines of at least moderate severity at maximum frown by investigator's assessment.
* Women of childbearing potential must have a negative serum pregnancy test at screening

Exclusion Criteria:

* Patients with an inability to substantially lessen glabellar lines by physically spreading them apart.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication
* Patients with an anaphylactic response history to botulinum toxin type A.
* Patients who have been administered botulinum toxin type A within the previous 6 months.
* Pregnant or lactating women.
* Participation in any research study involving drug administration within 90 days preceding enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-12-07 (Actual); Primary Completion 2012-03-30 (Actual); Study Completion 2012-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Foley, Doctor, Principal Investigator — Austrailia
Locations (1):
- Melbourne, Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- MT10109 A Unit: Single dose intramuscular injection of MT10109 (A Unit) at glabellar line (GL)
- MT10109 B Unit: Single dose intramuscular injection of MT10109 (B Unit) at glabellar line (GL)
- MT10109 C Unit: Single dose intramuscular injection of MT10109 (C Unit) at glabellar line (GL)
- Botox (Registered Trade Mark): Single dose intramuscular injection of Botox (B Unit) at glabellar line (GL)
Period: Overall Study
Arm/Group | MT10109 A Unit | MT10109 B Unit | MT10109 C Unit | Botox (Registered Trade Mark)
Started | 31 | 31 | 27 | 32
Completed | 28 | 23 | 25 | 26
Not Completed | 3 | 8 | 2 | 6

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- Total: Total of all reporting groups
Arm/Group | MT10109 A Unit | MT10109 B Unit | MT10109 C Unit | Botox (Registered Trade Mark) | Total
Number analyzed (Participants) | 31 | 31 | 27 | 32 | 121
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 44.9 (8.32) | 44.0 (9.77) | 45.3 (9.51) | 45.1 (9.53) | 44.8 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 24 | 27 | 107
  Male | 4 | 2 | 3 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 31 | 31 | 27 | 31 | 120
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 31 | 31 | 27 | 32 | 121

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Rating of Glabellar Line Severity at Maximum Frown by Live Assessment.
Description: Subjects included in the analysis had to have a baseline glabellar line (GL) severity rating at maximum frown of moderate (2) or severe (3). The GL severity were measured using a 4-point scale (0: none; 1: mild; 2: moderate; 3: Severe). A responder was defined as having a severity rating of none (0) or mild (1) at the corresponding post-baseline visit. Percentages are based on the number of subjects with an assessment at the relevant visit (Day 30).
Time Frame: at Day 30
Population: Full Analysis Set - comprised all randomized subjects who received at least one dose of study treatment and who had a glabellar lines severity rating at maximum frown at baseline and at least one post-baseline measurement.
Measure: Count of Participants; unit: Participants
Groups:
- MT0109 B Unit: Single dose intramuscular injection of MT10109 (B Unit) at glabellar line (GL)
Arm/Group | MT10109 A Unit | MT0109 B Unit | MT10109 C Unit | Botox (Registered Trade Mark)
Number analyzed (Participants) | 30 | 26 | 25 | 26
Participants
  Responders at Day 30 at Max Frown | 18 | 18 | 22 | 19
  Non-responders at Day 30 at Max Frown | 12 | 8 | 3 | 7

ADVERSE EVENTS:
Time Frame: Until the End-of-Study Visit (Day 120)
Description: This section focuses primarily on treatment-emergent adverse events (TEAEs), i.e., Adverse Events that started or worsened after the administration of study treatment.
Arm/Group | MT10109 A Unit | MT10109 B Unit | MT10109 C Unit | Botox (Registered Trade Mark)
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 1/27 | 1/32
Other Adverse Events (participants affected / at risk) | 7/31 | 7/31 | 10/27 | 10/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT10109 A Unit (N=31) | MT10109 B Unit (N=31) | MT10109 C Unit (N=27) | Botox (Registered Trade Mark) (N=32)
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT10109 A Unit (N=31) | MT10109 B Unit (N=31) | MT10109 C Unit (N=27) | Botox (Registered Trade Mark) (N=32)
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
NODULE (General disorders) | 0 | 1 | 0 | 0
ACUTE TONSILLITIS (Infections and infestations) | 0 | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 0
EYELID INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 0 | 3
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 1 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
HEAD DISCOMFORT (Nervous system disorders) | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 0 | 4
MIGRAINE (Nervous system disorders) | 0 | 1 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 1 | 0 | 0
TENSION HEADACHE (Nervous system disorders) | 0 | 1 | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 1 | 0 | 0
BREAST MASS (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
SEBACEOUS HYPERPLASIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less